CLINICAL TRIAL: NCT01052883
Title: A Phase I, Open Label, Randomized, Single Dose, Crossover Study in Healthy Subjects to Compare the Oral Bioavailability of a Prototype Tablet Formulation of Darunavir 800mg(G002) to That of the Commercial 400mg(F030) Tablet Formulation Under Fed & Fasted Conditions, in Presence of Low-dose Ritonavir
Brief Title: TMC114-TiDP3-C182 - A Study to Compare the Oral Bioavailability of a 800 mg Prototype Tablet Formulation of Darunivar (DRV) to That of the 400 mg Commercial Tablet Formulation in the Presence of Low Dose Ritonavir, Under Fasted and Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tibotec Pharmaceuticals, Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR016903
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2013-09

CONDITIONS: HIV Infections
Keywords: TMC114-TiDP3-C182; TMC114-C182; TMC114; HIV; HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Ritonavir

ARMS (4):
- 1 (Experimental): DRV commercial formulation/ DRV new formulation/ rtv 100mg tab DRV two 400 mg commercial formulation tablets in the morning of day 3 after food + rtv 100 mg 1/day on Day 1-5 [Treatment A] then after 7 days off treatment start DRV 800 mg new formulation tablet in the morning of Day 3 after food + rtv 100 mg 1/day on Day 1-5 [Treatment B]
  Interventions: Drug: DRV commercial formulation/ DRV new formulation/ rtv 100mg tab
- 2 (Experimental): DRV commercial formulation/ DRV new formulation/ rtv 100mg tab DRV 800 mg new formulation tablet/rtv 100mg tablet in the morning of Day 3 after food+ rtv 100 mg 1/day on Day 1-5 [Treatment B] then after 7 days off treatment start DRV two 400 mg commercial formulation tablets in the morning of day 3 after food + rtv 100 mg 1/day on Day 1-5 [Treatment A]
  Interventions: Drug: DRV commercial formulation/ DRV new formulation/ rtv 100mg tab
- 3 (Experimental): DRV commercial formulation/ DRV new formulation/ rtv 100mg tab DRV two 400 mg commercial formulation tablets in the morning of day 3 fasting + rtv 100 mg 1/day on Day 1-5 [Treatment C] then after 7 days off treatment start DRV 800 mg new formulation in the morning of day 3 fasting + rtv 100 mg 1/day on Day 1-5 [Treatment D]
  Interventions: Drug: DRV commercial formulation/ DRV new formulation/ rtv 100mg tab
- 4 (Experimental): DRV commercial formulation/ DRV new formulation/ rtv 100mg tab DRV 800 mg new formulation in the morning of day 3 fasting + rtv 100 mg 1/day on Day 1-5 [Treatment D] then after 7 days off treatment start DRV two 400 mg commercial formulation tablets in the morning of day 3 fasting + rtv 100 mg 1/day on Day 1-5 [Treatment C]
  Interventions: Drug: DRV commercial formulation/ DRV new formulation/ rtv 100mg tab

INTERVENTIONS:
Drug: DRV commercial formulation/ DRV new formulation/ rtv 100mg tab — DRV two 400 mg commercial formulation tablets in the morning of day 3 fasting + rtv 100 mg 1/day on Day 1-5 [Treatment C], then after 7 days off treatment start DRV 800 mg new formulation in the morning of day 3 fasting + rtv 100 mg 1/day on Day 1-5 [Treatment D]
  Arms: 3
Drug: DRV commercial formulation/ DRV new formulation/ rtv 100mg tab — DRV 800 mg new formulation tablet/rtv 100mg tablet in the morning of Day 3 after food+ rtv 100 mg 1/day on Day 1-5 [Treatment B], then after 7 days off treatment start DRV two 400 mg commercial formulation tablets in the morning of day 3 after food + rtv 100 mg 1/day on Day 1-5 [Treatment A]
  Arms: 2
Drug: DRV commercial formulation/ DRV new formulation/ rtv 100mg tab — DRV 800 mg new formulation in the morning of day 3 fasting + rtv 100 mg 1/day on Day 1-5 [Treatment D], then after 7 days off treatment start DRV two 400 mg commercial formulation tablets in the morning of day 3 fasting + rtv 100 mg 1/day on Day 1-5 [Treatment C]
  Arms: 4
Drug: DRV commercial formulation/ DRV new formulation/ rtv 100mg tab — DRV two 400 mg commercial formulation tablets in the morning of day 3 after food + rtv 100 mg 1/day on Day 1-5 [Treatment A], then after 7 days off treatment start DRV 800 mg new formulation tablet in the morning of Day 3 after food + rtv 100 mg 1/day on Day 1-5 [Treatment B]
  Arms: 1

SUMMARY:
The purpose of this study is to compare the drug levels of darunavir obtained after administration of a single administration of the 800 mg tablet (new formulation) to that following administration of two 400 mg commercial tablets formulation when administered under fed and fasted conditions to those also taking low-dose ritonavir. Darunavir is marketed for the treatment of HIV. The short-term safety and tolerability of darunavir following administration of a single 800 mg dose of darunavir given to healthy volunteers taking taking low-dose ritonavir will also be assessed.

DETAILED DESCRIPTION:
This is an open label study, which means that all parties including the study doctor, the healthy volunteer and the sponsor will know at all times which treatment group the volunteer is in. This is a cross over trial, which means that every volunteer will be sequentially subjected to 2 different treatments. A total of 32 healthy volunteers will participate in this study. Volunteers will be divided over 2 panels of 16 volunteers each. Volunteers in Panel 1 will be randomly assigned to treatment sequence AB or BA. Volunteers in Panel 2 will be randomly assigned to treatment sequence CD or DC. During all treatment periods 100 mg ritonavir (rtv) will be dosed once daily on Day 1 to Day 5. In treatment A you will receive a single dose of darunavir (DRV) two 400 mg commercial formulation in the morning of day 3 after a standard breakfast. In treatment B you will receive a single dose of darunavir (DRV) 800 mg new formulation in the morning of Day 3 also under fed conditions. In treatment C you will receive a single dose of darunavir (DRV) two 400 mg commercial formulation in the morning of day 3 under fasted conditions. In treatment D you will receive a single dose of darunavir (DRV) 800 mg new formulation in the morning of day 3 also under fasted conditions. Treatment sessions are organized with 7 days between treatment periods. In each session, an extensive investigation of the levels of DRV and rtv in the blood circulation is planned. Levels of DRV will be assessed at 15 different time points, i.e. before administration of DRV 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 12, 24, 48 and 72 hours after intake of DRV. Levels of rtv will be assessed at 13 different time points, i.e. before administration of rtv on Day 3, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9 and 12 hours after intake of rtv on day 3 and before administration of rtv on Day 4. Standard Safety assessments (blood biochemistry and hematology, urine analysis, ECG, pulse rate and blood pressure) will be performed on Day1, 3 and 6 in each Treatment period. Two 400 mg DRV commercial tablet formulation (F030) single dose on Day 3 of treatment A and C; 800 mg DRV new tablet formulation (G002) single dose on Day 3 of treatment B and D; 100 mg rtv capsule once daily on Day 1 to Day 5. All intake are oral.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking, or smoking no more than 10 cigarettes, or 2 cigars, or 2 pipes per day for at least 3 months prior to selection
* Normal weight as defined by a Body Mass Index (BMI, weight in kg divided by the square of height in meters) of 18.0 to 30.0 kg/m2, extremes included
* Use of effective non hormonal birth control methods, or willing to continue practicing these birth control methods for at least 30 days after the end of the treatment period for female volunteers of childbearing potential
* Negative serum pregnancy test and will not be breast feeding at screening
* Able to comply with protocol requirements
* Healthy on the basis of a medical evaluation that reveals the absence of any clinically relevant abnormality and includes a physical examination, medical history, electrocardiogram (ECG), vital signs, and the results of blood biochemistry, blood coagulation, and hematology tests and a urinalysis carried out at screening

Exclusion Criteria:

* Positive HIV 1 or HIV 2 test at screening
* Hepatitis A, B or C infection at screening
* History of significant skin disease such as, but not limited to rash or eruptions, food allergy or psoriasis
* Allergy, hypersensitivity or intolerance to DRV and rtv
* History of allergy to drugs such as, but not limited to, sulphonamides and penicillins

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Plasma levels of DRV 800 mg new formulation compared with 2x400 mg commercial formulation in fed and fasted conditions and in presence of low dose rtv | Plasma levels of DRV in each session at 15 timepoints and plasma levels of rtv after intake on Day 3 at 13 timepoints

SECONDARY OUTCOMES:
The short-term safety and tolerability of darunavir following administration of a single 800 mg dose of darunavir in the presence of low-dose ritonavir | 9 weeks (this includes treatment, washout and follow up period and is excluding screening period of maximum 21 days before first medication intake)

CONTACTS AND LOCATIONS:
Overall Officials: Tibotec Pharmaceuticals Clinical Trial, Study Director — Tibotec Pharmaceutical Limited

REFERENCES:
- [Derived] Kakuda TN, Leopold L, Timmers M, Van De Casteele T, Hillewaert V, Tomaka FL, Hoetelmans RM. Bioavailability and bioequivalence of a darunavir 800-mg tablet formulation compared with the 400-mg tablet formulation. Int J Clin Pharmacol Ther. 2014 Sep;52(9):805-16. doi: 10.5414/cp202066. PMID 25109510